CLINICAL TRIAL: NCT05277077
Title: The Effects of Pain Neuroscience Education Following Arthroscopic Rotator Cuff Repair on Clinical Outcomes
Brief Title: Pain Neuroscience Education Following Arthroscopic Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Caner Karartı, Caner Karartı, Hacettepe University, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022100
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Rotator Cuff Injuries; Tear; Pain, Shoulder
Keywords: Rotator Cuff Injuries; tear; pain; shoulder
MeSH Terms: conditions — Rotator Cuff Injuries; Lacerations; Shoulder Pain; Pain

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Investigator, Outcomes Assessor
Masking Description: the double blinded study (assessor and statistician)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): In addition to the conservative treatment, the experimental group will follow PNE sessions (one session per week over six consecutive weeks). Each session will take between 45 min and 1 h. The physiotherapist with 6 years of clinical and PNE experience will conduct all sessions. PNE will be conducted in line with international guidelines and covered the neurophysiology of pain, transition from acute to chronic pain, and the nervous system ability to modulate the pain experience. The theoretical information will be complemented with pictures and diagrams based on previous procedures. A booklet with the contents of each session and containing a mixture of text, figures, and activities to perform between sessions will be developed for the purpose of this study and given to participants. Time devoted to PNE will decrease from session 1 (60 min) to session 6 (15 min).
  Interventions: Other: Pain neuroscience education
- Control Group (Active Comparator): The control group will follow a conservative treatment. The 90-minute-long training sessions will be held 5 days per week. The training program will include the following exercises: cold-pack for 20 minutes; 20 minutes of Conventional TENS; 3 minutes of soft tissue massage for deltoid and biceps muscles; scapula and glenohumeral joint mobilizations; towel sliding and duster slide exercises on the wall; wand-assisted bilateral shoulder elevation; external rotation in increasing abduction angles, internal rotation in abduction, horizontal adduction and functional internal rotation exercises; strengthening exercises; finger ladder exercises; activation of deltoid, rotator cuff, and scapular muscles at chest level as the degree of active elevation increases; anterior elevation using an elastic band; strength training in "Full Can" position; closed kinetic chain trainings; isometric exercises of the periscapular muscles, deltoid and trapezius; and posterior capsule stretching.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Pain neuroscience education — The experimental group will follow a PNE protocol based on previous procedure for a whole period of 6 weeks in addition the conventional treatment.
  Arms: Experimental Group
Other: Conventional treatment — Patients from both groups will receive a conventional 6-week treatment programme (30 treatment sessions, five a week, for 90min duration).
  Arms: Control Group

SUMMARY:
Pain neuroscience education (PNE) aims to explain to patients the biological and physiological processes involved in a pain experience and, more importantly, defocus the issues associated with the anatomical structures. It has been demonstrated for musculoskeletal pain, PNE provides compelling evidence in reducing pain, disability, pain catastrophization, and limited physical movement. Rotator cuff tears (RCT) often lead to pain aggrevation, deterioration of patients' functioning and considerable economic burden for health care resources requiring consultations, physiotherapy, radiological examinations and surgery. Despite costly arthroscopic surgeries and long-term physiotherapy treatments, satisfactory results are scarce. The lack of satisfactory results at the end of all this effort suggests that some practices should be revised. Although PNE is likely to have beneficial effects on shoulder pathomechanics, to our knowledge, there is no randomized controlled research in the relevant literature investigating the effects of PNE in patients with an RCT. The present study aims to examine the effectiveness of PNE on clinical outcomes in a sample of patients with RCT.

DETAILED DESCRIPTION:
Therapeutic interventions based on pain neuroscience education (PNE) have emerged as promising. It consists of educational sessions describing the neurobiology and neurophysiology of chronic pain and pain processing, with a particular focus on the role of the central nervous system on chronic pain and deemphasizing anatomical issues. PNE promotes the patients' understanding of chronic pain and changes maladaptive thoughts and cognitions (e.g. pain catastrophizing), which are important barriers to active therapy and exercise. Despite the apparent complexity of neuroscience education, patients are able to understand and remember it. Furthermore, there is evidence that an educational strategy addressing neurophysiology and neurobiology of pain can have a positive effect on pain, disability, catastrophizing, and physical performance, especially if combined with exercise. Rotator cuff tears (RCT) often lead to pain aggrevation, deterioration of patients' functioning and considerable economic burden for health care resources requiring consultations, physiotherapy, radiological examinations and surgery. Despite costly arthroscopic surgeries and long-term physiotherapy treatments, satisfactory results are scarce. The lack of satisfactory results at the end of all this effort suggests that some practices should be revised. Although PNE is likely to have beneficial effects on shoulder pathomechanics, to our knowledge, there is no randomized controlled research in the relevant literature investigating the effects of PNE in patients with an RCT. The present study aims to examine the effectiveness of PNE on clinical outcomes in a sample of patients with RCT.

ELIGIBILITY:
Inclusion Criteria:

* being in the age range of 18-65 years
* being diagnosed with a small and medium-sized RCT based on magnetic resonance imaging and clinical continuity tests
* history of arthroscopic rotator cuff repair (ARCR)
* having a good command of the Turkish language
* scoring above 24 in the Mini Mental State Test
* ≥80% compliance in completing the post-ARCR Phase 1 trainings
* volunteering to participate in the study.

Exclusion Criteria:

* diabetes mellitus
* neurological problems
* cervical disc herniation
* visual, verbal, and/or cognitive defects (aphasia, unilateral neglect, etc.)
* osteoarthritis, rheumatoid arthritis or other systemic inflammatory problems
* hypermobility, trauma, and/or inflammation that could be a contraindication for mobilization
* former shoulder fractures on the affected side
* partial RCT
* former surgery on the affected side
* a history of adhesive capsulitis;
* traumatic shoulder instability (subluxation-dislocation)
* patients who are in stage 3 and above on the Goutallier classification system
* receiving a corticosteroid injection on the affected side within 6 weeks prior to diagnosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 6 weeks
  VAS is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
Shoulder Pain and Disability Index (SPADI) | 6 weeks
  The SPADI is a 13 item self-reported questionnaire assessing pain and functional status. Each item is measured on a 0-10 scale and a 0-100 score calculated. Higher scores represent greater levels of pain and disability. The SPADI has been shown to have good test-re-test reliability and be sensitive to change.
The Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH) | 6 weeks
  DASH questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100.

SECONDARY OUTCOMES:
Catastrophizing | 6 weeks
  Pain Catastrophizing Scale (PCS) will be used to evaluate the patient's feelings, thoughts, and emotions related to cognitive characteristics of pain. It is a self-administered questionnaire with 13 items and 3 subscales: helplessness, magnification, and rumination. A 5-point scale is used for each item, with higher values representing greater catastrophizing. The scores for each item are added to determine the subscales, and the total score is calculated by the summation of all items. The PCS scores range from 0 to 52 points.
Hospital Anxiety and Depression Scale (HADS) | 6 weeks
  HADS will be used to assess anxiety and depression. HADS consists of 7 items for anxiety and 7 for depression. The items are scored on a 4-point scale from 0 (not present) to 3 (considerable).
Tampa-Scale of Kinesiophobia (TSK) | 6 weeks
  Participants will be assessed with Tampa-Scale of Kinesiophobia (TSK) in terms of presence of kinesiophobia. The TSK is a 17-item scale that measures the somatic focus of patients (beliefs about underlying and serious medical problems), and activity avoidance (beliefs about (re) injury or increased pain). The TSK has moderate construct, concurrent and predictive validity, good internal consistency, and a moderate to good retest reliability. Patients scoring high on the TSK, above 37 points, are likely to have fear of movement.
12-Item Short-Form Health Survey (SF-12) | 6 weeks
  Participants will be assessed with 12-Item Short-Form Health Survey (SF-12) in terms of quality of life. It is a self-administered survey and two scores can be measured: the Physical Component and the Mental Component. In both, scores range from 0 to 100, with the highest scores associated with better levels of quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andias R, Neto M, Silva AG. The effects of pain neuroscience education and exercise on pain, muscle endurance, catastrophizing and anxiety in adolescents with chronic idiopathic neck pain: a school-based pilot, randomized and controlled study. Physiother Theory Pract. 2018 Sep;34(9):682-691. doi: 10.1080/09593985.2018.1423590. Epub 2018 Jan 10. PMID 29319386
- [Background] Malfliet A, Kregel J, Coppieters I, De Pauw R, Meeus M, Roussel N, Cagnie B, Danneels L, Nijs J. Effect of Pain Neuroscience Education Combined With Cognition-Targeted Motor Control Training on Chronic Spinal Pain: A Randomized Clinical Trial. JAMA Neurol. 2018 Jul 1;75(7):808-817. doi: 10.1001/jamaneurol.2018.0492. PMID 29710099
- [Background] Wijma AJ, van Wilgen CP, Meeus M, Nijs J. Clinical biopsychosocial physiotherapy assessment of patients with chronic pain: The first step in pain neuroscience education. Physiother Theory Pract. 2016 Jul;32(5):368-84. doi: 10.1080/09593985.2016.1194651. Epub 2016 Jun 28. PMID 27351769
- [Background] Louw A, Diener I, Butler DS, Puentedura EJ. The effect of neuroscience education on pain, disability, anxiety, and stress in chronic musculoskeletal pain. Arch Phys Med Rehabil. 2011 Dec;92(12):2041-56. doi: 10.1016/j.apmr.2011.07.198. PMID 22133255
- [Background] Wood L, Hendrick PA. A systematic review and meta-analysis of pain neuroscience education for chronic low back pain: Short-and long-term outcomes of pain and disability. Eur J Pain. 2019 Feb;23(2):234-249. doi: 10.1002/ejp.1314. Epub 2018 Oct 14. PMID 30178503
- [Background] Ryosa A, Laimi K, Aarimaa V, Lehtimaki K, Kukkonen J, Saltychev M. Surgery or conservative treatment for rotator cuff tear: a meta-analysis. Disabil Rehabil. 2017 Jul;39(14):1357-1363. doi: 10.1080/09638288.2016.1198431. Epub 2016 Jul 6. PMID 27385156